CLINICAL TRIAL: NCT02171546
Title: A Two-part Study to Determine the Relative Bioavailability of Dabigatran Etexilate 150 mg Bid (Capsules) With and Without 600 mg Quinidine Sulfate Tablets (Part 1) and to Measure the Effect of Quinidine as a Probe Inhibitor of P-glycoprotein on the Absorption of Fexofenadine, a Probe Substrate of P-glycoprotein (Part 2) in Healthy Male and Female Volunteers (an Open-label, Randomised, Two Times Two-way Crossover Study)
Brief Title: Relative Bioavailability of Dabigatran Etexilate Capsules With and Without Quinidine Sulfate Tablets and to Measure the Effect of Quinidine on the Absorption of Fexofenadine in Healthy Male and Female Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.75
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Quinidine; fexofenadine

ARMS (4):
- Dabigatran etexilate capsules (Active Comparator)
  Interventions: Drug: Dabigatran etexilate capsules
- Dabigatran etexilate capsules and quinidine sulfate tablets (Experimental)
  Interventions: Drug: Dabigatran etexilate capsules; Drug: Quinidine sulfate tablets
- Fexofenadine tablets (Active Comparator)
  Interventions: Drug: Fexofenadine tablets
- Fexofenadine and quinidine sulfate tablets (Experimental)
  Interventions: Drug: Quinidine sulfate tablets; Drug: Fexofenadine tablets

INTERVENTIONS:
Drug: Dabigatran etexilate capsules
  Arms: Dabigatran etexilate capsules; Dabigatran etexilate capsules and quinidine sulfate tablets
Drug: Quinidine sulfate tablets
  Arms: Dabigatran etexilate capsules and quinidine sulfate tablets; Fexofenadine and quinidine sulfate tablets
Drug: Fexofenadine tablets
  Arms: Fexofenadine and quinidine sulfate tablets; Fexofenadine tablets

SUMMARY:
Part 1: To investigate the effect of quinidine, a P-glycoprotein (P-gp) probe inhibitor on the bioavailability of dabigatran etexilate,

Part 2: To determine the effect of quinidine on the bioavailability of fexofenadine, a probe substrate for P-gp

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests ;
2. Age ≥18 and Age ≤55 years;
3. Body Mass Index (BMI) ≥18.5 and BMI <30 kg/m2;
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation;
5. If female of child-bearing potential, not be pregnant or breast feeding, nor plan to become pregnant for the duration of the study and for 2 months after receiving the last dose of study drug, and have a negative serum pregnancy test within 14 days of treatment, and prior to dosing;
6. Females of child-bearing potential willing to use adequate contraception, defined as the use of hormonal (oral, injectable or implantable) or barrier method contraceptives, intrauterine device and agree to use the same method of contraception for at least 2 months after drug administration. Women who have undergone a total hysterectomy, have a history of bilateral tubal ligation or are at least 2 years post-menopausal are not considered to be of child-bearing potential.

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance;
2. Any evidence of a clinically relevant concomitant disease;
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders;
4. Surgery of the gastrointestinal tract (except appendectomy);
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders;
6. History of relevant orthostatic hypotension, fainting spells or blackouts;
7. Chronic or relevant acute infections;
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients);
9. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial;
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial;
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial;
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day);
13. Inability to refrain from smoking on trial days;
14. Alcohol abuse (more than 60 g/day);
15. Drug abuse;
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial);
17. Excessive physical activities (within one week prior to administration or during the trial);
18. Any laboratory value outside the reference range that is of clinical relevance;
19. Inability to comply with dietary regimen of trial site;
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
21. A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
22. Taking drugs which are known P-gp inhibitors or inducers (verapamil, phenothiazine antipsychotics, erythromycin, antifungal drugs or St. John´s Wort) within the last 4 weeks before screening;
23. Chronic use of oral contraception containing ethinyl estradiol as the only method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of dabigatran in plasma at steady state over one dosing interval) | Before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00 and 12:00 hours after dosing on day 3
Cmax,ss (maximum concentration of dabigatran in plasma at steady state) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
AUC0-∞ (area under the concentration-time curve of fexofenadine in plasma over the time interval from 0 to infinity) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
Cmax (maximum measured concentration of fexofenadine in plasma) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1

SECONDARY OUTCOMES:
AUC0-tz,ss (area under the concentration-time curve of dabigatran in plasma from the time point 0 after the last dose at steady state to the last quantifiable dabigatran plasma concentration within the uniform dosing interval τ) | 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24 and 48 hours after dosing on day 3
tz,ss (time of last measurable concentration of dabigatran in plasma within the dosing interval τ at steady state) | 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24 and 48 hours after dosing on day 3
tmax,ss (time from last dosing to the maximum concentration of dabigatran in plasma at steady state) | 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24 and 48 hours after dosing on day 3
CL/Fss (apparent clearance of dabigatran in the plasma at steady state) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
Cmin,ss (minimum measured concentration of dabigatran in plasma at steady state) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
Cavg (average concentration of dabigatran at steady state) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
C10,2 (total dabigatran concentration 10 hours after the second dabigatran etexilate administration) | Day 2, 22 hours after the first dose on day 1
tmin,ss (time from last dosing to the minimum concentration of dabigatran in plasma at steady state over a uniform dosing interval τ) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
MRTpo,ss (mean residence time of dabigatran in the body at steady state after oral administration) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
Vz/Fss (apparent volume of distribution of dabigatran during the terminal phase λz at steady state following an extravascular administration) | Before dose on day 1, day 2, before dose, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on Day 3
Cmax (maximum measured concentration of quinidine in plasma) | Pre-dose, 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00, 11:00, 13:00, 25:00 and 49 hours after dosing
AUC0-∞ (area under the concentration-time curve of quinidine in plasma over the time interval from 0 to infinity) | Pre-dose, 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00, 11:00, 13:00, 25:00 and 49 hours after dosing
AUC0-tz (area under the concentration-time curve of fexofenadine in plasma from the time point 0 after the last dose to the last quantifiable analyte plasma concentration within the uniform dosing interval τ) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
tmax (time from last dosing to the maximum measured concentration of fexofenadine in plasma) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
t½ (terminal half-life of fexofenadine in plasma) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
MRTpo (mean residence time of fexofenadine in the body after p.o. administration) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
CL/F (apparent clearance of fexofenadine in plasma following extravascular administration) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
Vz/F (apparent volume of distribution of fexofenadine during the terminal phase λz following an extravascular dose) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 1
t½ (terminal half-life of dabigatran in plasma at steady state) | Before dose, 0:30, 1:00,1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 48:00 hours after dosing on day 3
Cpre,ss (pre-dose concentration of dabigatran in plasma immediately before administration of the following dose at steady state) | Before dose on day 3, day 4, and day 5